CLINICAL TRIAL: NCT02964819
Title: Influence of Interferential Current Therapy in the Treatment of Individuals With Shoulder Impact Syndrome: A Randomized, Placebo Controlled Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51675615.3.0000.5511
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise; Electric Stimulation Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- exercise group (Active Comparator): Manual cervical traction, Myofascial release of upper trapezius muscle, 3 sets of 1 minute;Sleeper's stretch, during 3 series of 30 seconds,Punch exercise, Knee push-up plus, Prone V-raise exercise (arms abducted at 120°), rotador cuff exercise (internal rotation), rotador cuff exercise (external rotation), Rotation on the wall using a ball (internal rotation), Rotation on the wall using a ball (external rotation).
  Interventions: Other: exercise
- exercise + Interferential current group (Experimental): Addition to the exercise protocol performed in the exercise group the interferential current. Four self-adhesive electrodes (8x5 cm), two upper and two lower ones (forming a square) will be placed around the center of the shoulder. The electrodes will be positioned crosswise, following the parameters: 4KHz (carrier frequency), 1/1 second (swing pattern), 100 Hz Frequency modulation amplitude (AMF), 50 Hz (sweep frequency), automatic vector mode, With intensity at the motor threshold of sensation, with duration of 50 minutes.
  Interventions: Other: exercise; Device: Interferential current therapy
- exercise + US group (Placebo Comparator): In addition to the exercise protocol performed in the exercise group, an ultrasound device will be used. The appliance will be used off, without any individual participant having knowledge. For this, the individual will be asked to position himself in the dorsal position on the stretcher, the therapist will perform the application of the transducer head, with gel on its surface, in the anterolateral region of the affected shoulder.
  Interventions: Other: exercise; Device: Therapeutic Ultrasound

INTERVENTIONS:
Other: exercise
Device: Interferential current therapy
  Arms: exercise + Interferential current group
Device: Therapeutic Ultrasound
  Arms: exercise + US group

SUMMARY:
This project will analyze the influence of interferential current therapy in an exercise program for individuals with a unilateral impact syndrome diagnosis. To that end, volunteers of both genders, aged 18-59 years, had an unilateral, unilateral pain in the shoulder with more than 3 months duration, at least grade 4 pain by the numerical scale of pain assessment, positivity In at least 2 of 3 orthopedic tests for impact syndrome, will be randomized into the following groups: exercise group, exercise + ultrasound group, exercise group + interferential current. Sixteen consecutive treatment sessions will be performed, and the volunteers will be evaluated before and after, by means of the following instruments: Numerical scale of evaluation of pain, Shoulder pain and disability index (SPADI), Pain-Related Catastrophizing Thoughts Scale, being applied the Numerical scale of evaluation of pain at the end of Each session and one month after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of anterolateral, unilateral pain in the shoulder with more than 3 months duration.
* Medical diagnosis,
* minimal grade 4 pain by numerical scale of pain assessment,
* positivity in at least 2 of 3 orthopedic tests for impact syndrome: Neer, Hawkins or Jobe.

Exclusion Criteria:

* Fibromyalgia diagnosis,
* pregnancy,
* numbness or tingling in the upper limb
* History of shoulder trauma, other shoulder related diseases,
* ruptured tendons, ligament laxity,
* symptoms of numbness and / or Tingling in the upper limbs, history of shoulder and / or cervical surgery
* use of corticosteroid injection in the shoulder, and analgesic, anti-inflammatory or muscle relaxant use and have or have undergone physiotherapeutic treatment in the last 6 months.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
physical function and pain | 10 months
  The Shoulder pain and disability index in the numerical version consists of 13 items distributed in the domain of pain (five items) and function (eight items), each item being scored on a numerical rating scale of 0 to 10 points. The final score of the questionnaire, as well as the score obtained separately by each domain, is converted into a percentage for values ranging from 0 to 100, with the highest score indicating worse shoulder dysfunction condition.

SECONDARY OUTCOMES:
pain | 10 months
  Numeric pain rating scale
Catastrophizing of the Pain | 10 months
  Pain-Related Catastrophizing Thoughts Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil